CLINICAL TRIAL: NCT03815331
Title: Xiaflex® Plus Testosterone Treatment Pilot Study Protocol A Six-month, Pilot Project of Testosterone Treatment in Subjects Who Are Undergoing Xiaflex® Therapy for the Treatment of Peyronie's Disease
Brief Title: Xiaflex® Plus Testosterone Treatment Pilot Study Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Men's Health Boston (Other)
Responsible Party: Principal Investigator, Dr. Abraham Morgentaler, PI/MD, Men's Health Boston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHB024
Record Dates: First submitted 2019-01-14; First posted 2019-01-24 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Peyronie's Disease (PD)
Keywords: Peyronie's disease; Hypogonadism
MeSH Terms: conditions — Penile Induration; Hypogonadism | interventions — Microbial Collagenase; Testosterone Propionate

STUDY DESIGN:
Intervention Model Description: All 20 subjects will receive Xiaflex® plus T treatment (Aveed®). Data collected from this pilot project will be analyzed and compared to historical data regarding treatment for PD using Xiaflex® only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD treatment with Xiaflex® plus Aveed (Experimental): Peyronie's Disease treatment with Xiaflex® and Aveed®. All 20 subjects will be treated with Xiaflex® and Aveed®. The data collected from this pilot project will be analyzed and compared to historical data regarding treatment for PD with Xiaflex® alone.
  Interventions: Drug: Xiaflex®; Drug: Aveed

INTERVENTIONS:
Drug: Xiaflex® — medication indicated for the treatment of adult men with Peyronie's disease with a palpable plaque and curvature deformity of at least 30 degrees at the start of therapy. Xiaflex belongs to a family of enzymes called collagenases. Collagenases are proteinases that hydrolyze collagen in its native triple helical conformation under physiological conditions, resulting in lysis of collagen deposits. The signs and symptoms of Peyronie's disease are caused by a collagen plaque. Injection of XIAFLEX into a Peyronie's plaque, which is comprised mostly of collagen, may result in enzymatic disruption of the plaque. Following this disruption of the plaque, penile curvature deformity and patient bother caused by Peyronie's disease are reduced
Drug: Aveed — Aveed® is an FDA-approved medication for treatment of hypogonadism (low testosterone). It is not approved for the treatment of Peyronie's Disease. Aveed® 750 mg/3mL injection will be placed intramuscularly at the beginning of study, at four weeks, at 10 weeks thereafter.

SUMMARY:
In this open-label, six-month, pilot study of men with Peyronie's disease there will be one subject group consisting of 20 subjects. All subjects will receive Xiaflex® plus testosterone (T) treatment (Aveed®). Males included in the study must be 18-70 years old; have a history of PD for more than six months; and have at two serum total testosterone level less than 350 ng/dL within 30 days prior to enrollment. The primary objective of this pilot study is to determine whether testosterone therapy offers increased efficacy of Xiaflex® (collagenase clostridium histolyticum) in subjects undergoing treatment for Peyronie's disease.

Endpoints will include reduction in degree of curvature and response to the PDQ questionnaire. Secondary objectives will be to assess men for change in plaque size, quality of life parameters, and sexual function. Data collected from this pilot study will be analyzed and compared to historical data regarding treatment for PD using Xiaflex® only. This pilot study will establish preliminary evidence needed to continue more in-depth research regarding Xiaflex® with T therapy and serve as a means to evaluate feasibility of a full-scale study.

DETAILED DESCRIPTION:
During this single-center pilot study, there will be one subject group consisting of men with Peyronie's disease and testosterone deficiency. Subject age range will be 18-70 years. Each subject will participate for approximately 6 months. All 20 subjects will receive Xiaflex® plus T treatment (Aveed®). Data collected from this pilot project will be analyzed and compared to historical data regarding treatment for PD using Xiaflex® only.

The eligibility criterion for 2 samples of total testosterone (<350ng/dL) or free testosterone (1.5 ng/dL analog assay or 100pg/mL calculated free testosterone) was chosen with the aim of demonstrating what the effect of testosterone treatment is on men that fall into the low range. The remainder of the inclusion and exclusion criteria are designed to select subjects for whom protocol treatment is considered appropriate. All relevant medical and non-medical conditions will be taken into consideration when deciding whether this protocol is suitable for a particular subject.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read, write, and understand English
2. Age greater than or equal to 18
3. Age less than or equal to 70
4. Identification of acquired penile curvature of greater than 30 degrees and less than 90 degrees associated with palpable penile plaque on physical examination at screening
5. Screening total testosterone of less than 350 ng/dL, twice withine 30 days of treatment
6. Screening free testosterone of less than 1.5ng/dL (analog assay) or 100pg/mL (calculated)
7. Planning to initiate Xiaflex® injections at MHB
8. Willingness to initiate testosterone therapy
9. Willing to be followed at MHB for the next 3 months
10. Willing to provide informed consent for this study

Exclusion Criteria:

1. Prior history of treatment for PD that includes surgery
2. Prior treatment with oral therapy for PD unless at least stopped 2 weeks prior to signing the informed consent (e.g. Potaba, Vitamin E, colchicines)
3. Previous exposure to exogenous T, clomiphene citrate, or other Selective Estrogen Receptor Modulators, unless off therapy for at least 12 weeks
4. Presence of dense calcified plaque by ultrasound at screening
5. Hypersensitivity to testosterone, stearic acid, or polyvinylpyrolidone (the constituents of Aveed®)
6. Unwillingness to start testosterone therapy
7. Screening total testosterone of greater than 350 ng/dL
8. Screening free testosterone of more than 1.5ng/dL (analog assay) or 100pg/mL (calculated)
9. Unable to achieve adequate erection with penile injection to assess degree of curvature
10. Prior history of definitive treatment for prostate cancer, bladder cancer, or other pelvic malignancies including surgery, external beam radiation therapy, brachytherapy, cryotherapy
11. Prior history of prostate cancer, hematologic disorders, chronic liver disease including cirrhosis and hepatitis C, disorders affecting the immune system, including infection with human immunodeficiency virus, or psychiatric disorders including major depression, schizophrenia, bipolar disease
12. Prior history of cerebrovascular accident, history of deep venous thrombosis within the past 5 years or history of untreated or severe sleep apnea
13. Screening PSA more than 4.0 ng/mL, unless prostate cancer has been excluded to the Investigator's satisfaction
14. Incapable of giving informed consent or complying with the protocol

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
change in penile curvature | 6 months
  The primary objective of this study is to determine whether supplemental testosterone treatment offers change in efficacy to Xiaflex® (collagenase clostridium histolyticum) alone in selected men undergoing treatment for Peyronie's disease. The primary endpoints are change in degrees of penile curvature from baseline.
change in PDQ responses | 6 months
  change in global sexual satisfaction, as measured by the Peyronie's Disease Questionnaire (PDQ).
  Not a scale but direct comparison of patients sexual activity through patients' answers.

SECONDARY OUTCOMES:
Change in plaque size | 6 months
  (mm longest diameter)
Change in quality of life | 6 months
  (Patient Health Questionnaire) Scale total can range from 0 to 27 (Not difficult at all to very difficult) Higher values would be worse outcome
Quality of erections and satisfaction with sexual function | 6 months
  (International Index of Erectile Function) No scale, direct comparison of answers
Change in quality of life | 6 months
  (Low T Questionnaire) Scale total ranges from 0 to 84 (strongly agree to strongly disagree) Higher values would be worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Morgentaler, MD, Principal Investigator — Men's Health Boston
Locations (1):
- Men's Health Boston, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brock G, Hsu GL, Nunes L, von Heyden B, Lue TF. The anatomy of the tunica albuginea in the normal penis and Peyronie's disease. J Urol. 1997 Jan;157(1):276-81. PMID 8976279
- [Background] Moreno SA, Morgentaler A. Testosterone deficiency and Peyronie's disease: pilot data suggesting a significant relationship. J Sex Med. 2009 Jun;6(6):1729-1735. doi: 10.1111/j.1743-6109.2009.01250.x. Epub 2009 Mar 30. PMID 19473459
- [Background] Gonzalez-Cadavid NF, Magee TR, Ferrini M, Qian A, Vernet D, Rajfer J. Gene expression in Peyronie's disease. Int J Impot Res. 2002 Oct;14(5):361-74. doi: 10.1038/sj.ijir.3900873. PMID 12454687
- [Background] Devine CJ Jr, Somers KD, Jordan SG, Schlossberg SM. Proposal: trauma as the cause of the Peyronie's lesion. J Urol. 1997 Jan;157(1):285-90. doi: 10.1016/s0022-5347(01)65361-8. PMID 8976281
- [Background] Shen ZJ, Zhou XL, Lu YL, Chen ZD. Effect of androgen deprivation on penile ultrastructure. Asian J Androl. 2003 Mar;5(1):33-6. PMID 12647000
- [Background] Demling RH. The role of anabolic hormones for wound healing in catabolic states. J Burns Wounds. 2005 Jan 17;4:e2. PMID 16921407
- [Background] Hetzler LE, Sharma N, Tanzer L, Wurster RD, Leonetti J, Marzo SJ, Jones KJ, Foecking EM. Accelerating functional recovery after rat facial nerve injury: Effects of gonadal steroids and electrical stimulation. Otolaryngol Head Neck Surg. 2008 Jul;139(1):62-7. doi: 10.1016/j.otohns.2008.02.006. PMID 18585563
- [Background] Maus U, Andereya S, Schmidt H, Zombory G, Gravius S, Ohnsorge JA, Niedhart C. [Therapy effects of testosterone on the recovery of bone defects]. Z Orthop Unfall. 2008 Jan-Feb;146(1):59-63. doi: 10.1055/s-2007-989436. German. PMID 18324583
- [Background] Cavallini G, Biagiotti G, Lo Giudice C. Association between Peyronie disease and low serum testosterone levels: detection and therapeutic considerations. J Androl. 2012 May-Jun;33(3):381-8. doi: 10.2164/jandrol.111.012948. Epub 2011 Jun 30. PMID 21719695
- [Background] Stallard N. Optimal sample sizes for phase II clinical trials and pilot studies. Stat Med. 2012 May 20;31(11-12):1031-42. doi: 10.1002/sim.4357. Epub 2011 Nov 3. PMID 22052407
- [Result] Taylor FL, Levine LA. Peyronie's Disease. Urol Clin North Am. 2007 Nov;34(4):517-34, vi. doi: 10.1016/j.ucl.2007.08.017. PMID 17983892